CLINICAL TRIAL: NCT04432987
Title: Determination of Dornase Alpha Effectiveness in COVID-19 Treatment
Brief Title: Dornase Alpha for the Treatment of COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8820
Record Dates: First submitted 2020-06-15; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: COVID-19, Dornase Alpha
MeSH Terms: conditions — COVID-19 | interventions — dornase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Newly Diagnosed Patient Group (n=30) (Experimental): I. Dornase Alpha treated group (n=15)
  ii. Control group (n=15)
  Interventions: Drug: Pulmozyme
- Patient Group Monitored by Mechanical Ventilation (n=30) (Experimental): I. Dornase Alpha treated group (n=15)
  ii. Control group (n=15)
  Interventions: Drug: Pulmozyme

INTERVENTIONS:
Drug: Pulmozyme — PULMOZYME contains an active substance called dornase alpha as an active substance. Dornase alpha is a human-made version of a protein called DNase in your body and is also known as recombinant human deoxyribonuclease 1 or rhDNase.
  Drug will be administered at a dose of 2,5 mg/2 times per day for 7 days

SUMMARY:
In this study, the effectiveness of the Dornase Alpha treatment, which is known to reduce the viscosity of respiratory secretions, will be investigated in new diagnosed and severe COVID-19 patients separately.

DETAILED DESCRIPTION:
Recent studies confirmed the role of immune hyperactivation in the pathogenesis of COVID-19. Immune cells, especially neutrophils, infiltrate pulmonary capillaries that cause acute fibrin deposition and extravasation into the alveolar space. This excessive accumulation of neutrophils constitutes NETs which makes the mucus thick and viscous. The highly viscous mucus lowers the patient's respiratory function and impairs ventilation supporting NETs may play a major role in the disease. As a mechanism, double-stranded DNA constitutes the backbone of NETs and Dornase alfa promotes the clearance of NETs from plasma neutralization. Endogenous Deoxyribonucleases (DNases), which physiologically break up this extracellular DNA, may become overwhelmed by a massive influx of NETs. Clinically, recombinant human DNase I (rhDNase, Dornase Alfa) has the identical primary amino acid sequence with the native human enzyme and has been approved for the management of cystic fibrosis. Daily administration of dornase alfa is effective in the treatment of cystic fibrosis patients improving pulmonary functions. The similarity of mucus secretions in COVID-19 and cystic fibrosis patients by the means of NETs makes Dornase alfa as a therapeutic option in COVID-19.

Progressive COVID-19 pneumonia may be mortal if it is not treated early, causing respiratory failure. The most important factor leading to respiratory failure is hyaline membrane formed by a neutrophil trap that develops in the cavities of the alveoli. Dornase Alpha is thought to have an important contribution by the lysis of this hyalen membrane. In this study, it is aimed to evaluate the effectiveness of Dornase Alpha treatment in case of early and late use in COVID-19 disease.

Patients diagnosed with COVID-19 PCR and / or radiological-clinical findings is included in the study, and this treatment is carried out in 2 patient groups in comparison with the control groups. The groups are:

1. Newly Diagnosed Patient Group I. Dornase Alpha treated group ii. Control group
2. Patient Group Monitored by Mechanical Ventilation I. Dornase Alpha treated group ii. Control group

ELIGIBILITY:
Inclusion Criteria:

* Being 18 or older
* Approving the Informed Consent Form
* Being diagnosed with COVID-19 with PCR and / or radiological clinical findings
* Hospitalization indication according to Ministry of Health criteria

Exclusion Criteria:

* Pregnant and / or breastfeeding women.
* Any known allergy to Dornase Alpha
* Being involved in another drug study
* Previously diagnosed with chronic lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-08-25 (Estimated); Study Completion 2020-09-25 (Estimated)

PRIMARY OUTCOMES:
Response | 3 months
  i. The patient has no complaints (cough and dyspnea completely disappear, the number of breaths are in the age-appropriate range, oxygen saturation is in the normal range), inflammatory markers in blood improve (CRP, LDH, Ferritin and D-Dimer regression to the reference range).
  ii. Extubation (for mechanically ventilated group)
  iii. Intubated (for newly diagnosed group)

SECONDARY OUTCOMES:
Survival | 3 months
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Ercument Ovalı, MD, Principal Investigator — Acıbadem Labcell Cellular Therapy Laboratories
Locations (1):
- Acıbadem Altunizade Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No